CLINICAL TRIAL: NCT07353489
Title: Evaluation of the Safety and Efficacy of Single Use Powered Endoscopic Staplers and Cartridges in Thoracic Surgery: A Retrospective Clinical Study
Brief Title: easyEndoTM Powered in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-Elite-01
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- easyEndoTM Powered Single Use Powered Endoscopic Staplers and Cartridges (Experimental)
  Interventions: Device: easyEndoTM Powered Single Use Powered Endoscopic Staplers and Cartridges

INTERVENTIONS:
Device: easyEndoTM Powered Single Use Powered Endoscopic Staplers and Cartridges — Using easyEndoTM Powered Single Use Powered Endoscopic Staplers and Cartridges transection, resection, and/or creation of anastomoses in thoracic surgery

SUMMARY:
The goal of this retrospective, single-arm is to evaluate the safety and performance of the easyEndo™ Powered Single Use Powered Endoscopic Staplers and Cartridges in thoracic surgery. The main question it aims to answer is the safety and performance of the staplers

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent thoracic surgery (including lobectomy, segmentectomy, wedge resection, etc.) using easyEndo™ Powered Single-Use Powered Endoscopic Staplers and Cartridges at our hospital.
* Surgery date was on or after January 1, 2024.
* Patients with complete medical records (including demographic data, surgical details, perioperative management, and follow-up information).
* Patients who completed a 1-year postoperative follow-up, with available and valid follow-up data

Exclusion Criteria:

* Patients who used other brands or types of endoscopic staplers instead of easyEndo™ Powered Single-Use Powered Endoscopic Staplers and Cartridges during surgery.
* Surgery date was before January 1, 2024.
* Patients with incomplete medical records or missing key information (e.g., unclear surgical procedures, unrecorded stapler use details, lost to follow-up before 1 year).
* Patients with severe underlying diseases that may affect postoperative outcomes or follow-up, such as end-stage heart, liver, or kidney disease, severe coagulation disorders, or uncontrolled malignant tumors (other than the primary disease requiring thoracic surgery).
* Patients with allergies to the materials of easyEndo™ staplers or cartridges, or who experienced adverse reactions related to stapler material allergies intraoperatively or postoperatively.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
stapling success rate | Perioperative/Periprocedural
  no leakage intra-operation and post-operation

SECONDARY OUTCOMES:
Intraoperative blood loss volume | Perioperative/Periprocedural
Blood transfusion requirement | Perioperative/Periprocedural
Conversion to open thoracotomy | Perioperative/Periprocedural
Length of hospital stay | Perioperative/Periprocedural
Postoperative drainage duration | Perioperative/Periprocedural
total drainage volume | Perioperative/Periprocedural
Reoperation requirement | Perioperative/Periprocedural
The incidence of complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jining Medical University, Jining, Shandong, China

IPD SHARING:
Plan to Share IPD: No